CLINICAL TRIAL: NCT00124891
Title: Study Evaluating Subjects With Non-sustained Ventricular Tachycardia
Brief Title: Study Evaluating GAP-486 in Non-sustained Ventricular Tachycardia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3163K1-200
Record Dates: First submitted 2005-07-13; First posted 2005-07-28 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Arrhythmias
Keywords: Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

INTERVENTIONS:
Drug: Double-blind investigational anti-arrhythmic
Drug: GAP-486

SUMMARY:
To determine whether the administration of test article will decrease the occurrence of ventricular arrhythmias in patients who have acute coronary syndrome (unstable angina, ST segment elevated myocardial infarction or myocardial infarction without ST elevation).

ELIGIBILITY:
INCLUSION CRITERIA:

* Male and female patients, 18 years of age or older, that have experienced an acute ischemic event within 24 hours prior to study entry.
* Patients with a documented history of coronary artery disease or left ventricular dysfunction
* Patients who have experienced an episode of non-sustained ventricular tachycardia within 24 hours of the index ischemic event

EXCLUSION CRITERIA:

* Patients who have had percutaneous coronary intervention (PCI), thrombolytics, or open-heart surgery within 48 hours prior to study entry, or who require it during test article administration
* Patients who have taken another antiarrhythmic medication (other than a beta blocker) within 5 half-lives of the start of test article
* Patients who have a history of torsades de pointes, long QT syndrome, QTc > 0.50

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2005-06-01 (Actual); Primary Completion 2006-11-01 (Actual); Study Completion 2006-11-01 (Actual)

PRIMARY OUTCOMES:
The total number of ventricular beats recorded by Holter monitoring during the 24 hr. on-therapy phase.

SECONDARY OUTCOMES:
The total number of NSVT beats, PVCs/couplets, NSVT episodes during the 24 hr. on-therapy phase and incidence of new-onset atrial fibrillation during the 24hr. on-therapy phase.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Brazil, xavierl@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Romania and Russia, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Mexico, gomezlj@wyeth.com; Trial Manager, Principal Investigator — For Italy, decresg@wyeth.com; Trial Manager, Principal Investigator — For Hungary, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For United Kingdom, ukmedinfo@wyeth.com; Trial Manager, Principal Investigator — For Sweden and Denmark, MedInfoNord@wyeth.com
Locations (60):
- United States (6):
  - Merced, California
  - Melbourne, Florida
  - Orlando, Florida
  - Peoria, Illinois
  - Iowa City, Iowa
  - Norfolk, Virginia
- Brazil (5):
  - Curitiba, Paraná
  - Porto Alegre, Rio Grande do Sul
  - São José, Rio Preto
  - São Paulo, São Paulo
  - Salvador
- Canada (10):
  - Calgary, Alberta
  - Surrey, British Columbia
  - Newmarket, Ontario
  - Oshawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Saint-Hyacinthe, Quebec
  - Sherbrooke, Quebec
  - Terrebonne, Quebec
  - Moose Jaw, Saskatchewan
- Multiple Locations, Croatia
- Denmark (3):
  - Copenhagen
  - Copenhagen South
  - Frederiksberg
- Hungary (4):
  - Tószegi U. 21., H-5004 Szolnok
  - Nyíri U. 38., H-6000 Kecskemét
  - Markusovszky U. 3., H-9700 Szombathely
  - Seregélyesi, Székesfehérvár
- India (6):
  - Hyderabad, Andhra Pradesh
  - Thellakom, Kottayam
  - Bandra, Mumbai
  - Multiple Locations, New Delhi
  - Rajasthan, Rajasthan
  - Multiple Locations
- Italy (4):
  - Multiple Locations, Pisa
  - Genova
  - Multiple Locations
  - Roma
- Mexico (7):
  - México, D.F.
  - Libertad, Guadalajara Jalisco
  - Multiple Locations, Guadalajara Jalisco
  - Zapopan, Guadalajara Jalisco
  - Monterrey, Nuevo León
  - Padilla, Veracruz
  - Tlalpan
- Poland (3):
  - Ostrowiec Świętokrzyski
  - Piotrkow Trybunalski
  - Warsaw
- Bucharest, Romania
- Russia (2):
  - Moscow
  - Saint Petersburg
- Serbia (2):
  - Belgrade
  - Kamenitz
- Gothenburg, Sweden
- Ukraine (3):
  - Kiev
  - Kyiv
  - Odesa
- United Kingdom (2):
  - Newcastle upon Tyne
  - Nottingham